CLINICAL TRIAL: NCT03087526
Title: Non Invasive Prenatal Diagnosis on Isolated Circulating Fetal Trophoblastic Cells (CFTC) for Triplet Repeat Diseases
Brief Title: NIPD on CFTC for Triplet Repeat Diseases
Acronym: DIACCIMEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL17_0021
Record Dates: First submitted 2017-02-23; First posted 2017-03-22 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Non Invasive Prenatal Diagnosis
Keywords: Non Invasive Prenatal Diagnosis (NIPD); Circulating Fetal Trophoblastic Cells (CFTC); Huntington's Disease; Myotonic Dystrophy Type 1; Fragile X syndrome; Spinocerebellar Ataxia type 1; Spinocerebellar Ataxia type 2; Spinocerebellar Ataxia type 3
MeSH Terms: conditions — Huntington Disease; Myotonic Dystrophy; Fragile X Syndrome; Spinocerebellar Ataxias; Machado-Joseph Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Couple at risk of transmitting a triplet-repeat disease (Experimental): Expectant couple (pregnant woman between 9 and 34 weeks of gestation and her spouse) at risk of transmitting a triplet-repeat related genetic disease among Huntington disease, Myotonic Dystrophy type 1, Fragile X syndrome, Spinocerebellar Ataxia type 1, Spinocerebellar Ataxia type 2, Spinocerebellar Ataxia type 3
  Interventions: Genetic: Non invasive prenatal diagnosis

INTERVENTIONS:
Genetic: Non invasive prenatal diagnosis — Search for the familial mutation on isolated circulating fetal trophoblastic cells from maternal blood

SUMMARY:
The purpose of this study is to develop and validate an analytical and clinical NIPD test for triplet repeat diseases by isolated circulating fetal trophoblastic cells (CFTC) analysis from maternal blood, searching for the familial mutation in families at risk of having one of the following triplet repeat diseases: Huntington's disease, Steinert Myotonic dystrophy, Fragile X syndrome, spinocerebellar ataxia (SCA) 1, 2 and 3.

DETAILED DESCRIPTION:
Non Invasive Prenatal Diagnosis (NIPD), based on the analysis of circulating cell-free fetal DNA (cff-DNA) is very promising for early diagnosis of monogenic diseases. Such an approach is a safer alternative to invasive methods of prenatal testing (amniocentesis or choriocentesis) which entails a significant risk of miscarriage (0.5%-1%). However, technical issues related to the characteristics of cff-DNA remain and do not allow the search of all the mutations, in particular triplet expansion mutations which concern rare and incurable diseases (Huntington's disease, Steinert Myotonic dystrophy, Fragile X syndrome, SCA1, 2, 3). Indeed, the strong fragmentation and the short size of cff-DNA (143 bp) do not allow direct detection of these mutations. However, Prenatal Diagnosis (PND) requests for this group of pathologies represent the second most frequent PND indication at the national level after cystic fibrosis (ABM 2013). An alternative approach is to perform analysis on circulating fetal trophoblastic cells (CFTC) from maternal blood. Several methods have been used to isolate CFTCs from maternal blood. However, to date, no test is reliable enough for a routine application to replace invasive protocols. Recently, new enrichment systems have been optimized for circulating tumor cells (CTCs) as a liquid biopsy of cancer. Some of these new technologies can be easily applied to the isolation and characterization of CFTCs. The objective of this study is to complete our NIPD services by developing an approach on CFTC adapted to the analysis of triplet repeat diseases, which cannot be performed on cff-DNA.

It is a multicenter, prospective study for performance evaluation of a diagnostic method. The subjects included will be pregnant women between 9 and 34 weeks of gestation and their partner (future fathers). Pregnant woman and future father genotypes (sick or healthy) are known for one of the following diseases: Huntington's disease, Steinert's myotonic dystrophy, fragile X and spinocerebellar ataxias types 1, 2 or 3. The main objective is achieved by the agreement between gold standard (PND by amniocentesis or choriocentesis) and NIPD results for each pregnant woman participating in the study (the absence or presence of the mutated allele).

The couple inclusion will take place in one of the participating medical genetic centers during genetic counseling consultation for a pregnancy at risk for one of the pathologies mentioned above.

During this visit, the pregnant woman's blood sample (blood sample taken on 3 x 10 ml BCT and 5 ml on EDTA) and the future father (5 ml on EDTA) will be carried out. The duration of inclusion is the time of the visit. Blood collection of pregnant women on cell-free DNA "Blood Collection Tubes" (BCT) to screen CFTCs will be addressed to the Human Rare Circulating Cells Laboratory (LCCRH). The molecular analysis of the CFTC isolated by the LCCRH as well as the genomic DNA extraction and analysis (from the 5 ml of blood on EDTA) of the couple will be carried out by the Laboratory of Molecular Genetics (LGM) located in the same Building (IURC - Montpellier University Hospital).

The analysis performed on a simple maternal blood test will allow to determine whether the future child is affected or not by the inherited disease. With this new NIPD approach, there could be a 50% decrease in the use of the invasive method for PND. This analysis can be offered to women carrying foetuses at risk for triplet repeat diseases. Finally, this approach can be applied to any monogenic diseases by CFTCs isolation automation from maternal blood.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years old
* pregnant woman between 9 and 34 weeks of gestation
* Couple at risk (based on family history or echographic findings) for one of the following diseases: Huntington's disease, Steinert's myotonic dystrophy, fragile X and spinocerebellar ataxias 1, 2 or 3
* Written informed consent was obtained for the study
* Prenatal diagnosis has been programmed for the current pregnancy during which maternal blood is collected
* Couple molecular diagnosis results for one of the following diseases (Huntington's disease, Steinert's myotonic dystrophy, fragile X and spinocerebellar ataxias 1, 2 or 3 ) MUST BE AVAILABLE.

Exclusion Criteria:

* Couple Genomic DNA are unavailable
* Subjects at risk of transmitting the family disease, but not wishing to know their molecular status
* individuals under guardianship by court order

Min Age: 18 Months | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Concordance rate between cell-based genetic non invasive prenatal test and gold standard prenatal test (choriocentesis or amniocentesis). | 30 months
  Analysis of the concordance of the prenatal results obtained by our new NIPD (Non-Invasive Prenatal Diagnosis) approach and those blindly obtained during the gold-standard prenatal genetic test will be carried out for each pregnant woman participating in the study.

SECONDARY OUTCOMES:
Non Invasive Prenatal Diagnostic test failure rate. | 30 months
  Count of the women enrolled for whom NIPD test will be inconclusive (because of insufficient circulating fetal cells isolation or allele drop out making accurate haplotyping impossible).

CONTACTS AND LOCATIONS:
Overall Officials: Marie Claire VINCENT, PhD-PharmaD, Principal Investigator — University Hospital, Montpellier
Locations (8):
- France (8):
  - CHU Bordeaux, Bordeaux
  - CHU Montpellier, Montpellier
  - CHU Nice, Nice
  - CHU Nîmes, Nîmes
  - CHU Rennes, Rennes
  - CH Saint Brieuc, Saint-Brieuc
  - CHU Strasbourg, Schiltigheim
  - CHU Toulouse, Toulouse

REFERENCES:
- [Result] Cayrefourcq L, Vincent MC, Pierredon S, Moutou C, Imbert-Bouteille M, Haquet E, Puechberty J, Willems M, Liautard-Haag C, Molinari N, Zordan C, Dorian V, Rooryck-Thambo C, Goizet C, Chaussenot A, Rouzier C, Boureau-Wirth A, Monteil L, Calvas P, Miry C, Favre R, Petrov Y, Khau Van Kien P, Le Boette E, Fradin M, Alix-Panabieres C, Guissart C. Single Circulating Fetal Trophoblastic Cells Eligible for Non Invasive Prenatal Diagnosis: the Exception Rather than the Rule. Sci Rep. 2020 Jun 17;10(1):9861. doi: 10.1038/s41598-020-66923-9. PMID 32555262
- [Result] Liautard-Haag C, Durif G, VanGoethem C, Baux D, Louis A, Cayrefourcq L, Lamairia M, Willems M, Zordan C, Dorian V, Rooryck C, Goizet C, Chaussenot A, Monteil L, Calvas P, Miry C, Favre R, Le Boette E, Fradin M, Roux AF, Cossee M, Koenig M, Alix-Panabiere C, Guissart C, Vincent MC. Noninvasive prenatal diagnosis of genetic diseases induced by triplet repeat expansion by linked read haplotyping and Bayesian approach. Sci Rep. 2022 Jul 6;12(1):11423. doi: 10.1038/s41598-022-15307-2. PMID 35794169